CLINICAL TRIAL: NCT04253301
Title: Feasibility of the InnoVein Valve and Delivery System for Chronic Venous Insufficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnoVein (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-CP-2001
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects will have the InnoVein Valve implanted
  Interventions: Device: InnoVein Valve Treatment

INTERVENTIONS:
Device: InnoVein Valve Treatment — Subjects will have the InnoVein Valve implanted

SUMMARY:
This objective of this feasibility study is to evaluate the safety of the InnoVein Valve and Delivery System for treatment of chronic venous insufficiency.

DETAILED DESCRIPTION:
Chronic Venous Insufficiency occurs when the venous wall and/or valves in the leg veins are not working effectively, making it difficult for blood to return to the heart from the legs.The core etiology of the disease stems from increased venous pressure and incompetent venous valves leading to regurgitation of blood that accumulates in the legs. It has been shown that implantation or recreation of a functional valve can lead to clearance of excess blood and resolution of symptoms.

The InnoVein Valve and Delivery System is a new, investigational biocompatible valve intended to support natural flow in vessels in patients with Chronic Venous Insufficiency. The purpose of this study is to assess the safety of the InnoVein Valve and Delivery System for treatment of Chronic Venous Insufficiency.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written Informed Consent
* Diagnosis of symptomatic non-obstructive chronic valvular insufficiency of the femoral vein
* Willing and medically able to receive intraprocedural and post-procedural anticoagulation medication
* Life expectancy >1yr
* Reflux time >1s in the superficial femoral and/or popliteal vein

Key Exclusion Criteria:

* Any prior deep vein intervention within 6 months prior to the Index Procedure
* History of 2+ DVTs
* Inadequate inflow to the femoral vein or inadequate outflow through the femoral vein, iliac vein, or IVC
* Current IVC Placement
* History of pulmonary embolism within 6 months
* Conditions that increase the risk of device thrombosis or patient bleeding
* Any planned surgical or interventional procedure within 30 days prior to or after the Index Procedure
* Investigator or sponsor believes the subject would not benefit, would not be appropriate, be unable to follow-up, or be at high risk for non-compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Safety of the InnoVein Valve and Delivery System: Number of Major Adverse Events | 30 Days
  Number of Major Adverse Events

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Flinders, Adelaide

IPD SHARING:
Plan to Share IPD: No